CLINICAL TRIAL: NCT03244345
Title: Depression, Stress and Vulnerability Factors in Drug Resistant Focal Epilepsies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-19; 2016-A00708-43 (Other: IDRCB)
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Depression and Epilepsy
MeSH Terms: conditions — Depression; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epileptic patient (Experimental)
  Interventions: Behavioral: Self-measurement scale of sensitivity to stress/emotion

INTERVENTIONS:
Behavioral: Self-measurement scale of sensitivity to stress/emotion — Patient will answer self-questionner on Depression

SUMMARY:
Psychiatric disturbances, notably depression, occur frequently as co-morbid conditions with epilepsy. A complex, probably bidirectional relationship between epilepsy and depression has been postulated. Both epilepsy and depression also interact with stressful life events, but only some patients develop these disorders after a stressful event, indicating the possibility of a "vulnerable" population. Animal and human studies have looked at the role of brain derived neurotrophic factor (BDNF) in this context. Low serum and/or CSF levels of BDNF are associated with higher incidence of depression, and thus indicate the vulnerable population.

Animal studies of BDNF have looked specifically at the relation between epilepsy and depression using a novel "double hit" design. After chronic stress exposure, measurement of BDNF levels allowed identification of 2 sub-groups: a vulnerable population and non-vulnerable population. A "second hit" of kainic acid induced status epilepticus (SE) was then applied to both the vulnerable and non-vulnerable populations. Only the vulnerable population exposed to SE developed a depression-like profile.

In a proof of concept approach we propose studying the relation between epilepsy, depression, anxiety and stressful life events, using serum BDNF levels in patients with pharmacoresistant epilepsy. Evaluation of epilepsy type and co-morbid psychiatric profile will be performed in 150 subjects. By comparing BDNF levels for different epilepsy subgroups to BDNF levels for healthy subjects and for depressed subjects without epilepsy, we hope to identify whether risk of co-morbid depression and/or anxiety in epilepsy may be predicted using BDNF levels. In addition, in a subgroup of 25 patients, we propose a pilot study in which cortisol and C-reactive protein will be measured in addition to BDNF.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of epilepsy, of any type (partial or generalised) and at any stage from diagnosis onwards
* Known or unknown etiology (symptomatic or cryptogenic epilepsy)

Exclusion Criteria:

* Psychogenic non-epileptic seizures
* Psychotic disorders and bipolar disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Depression | 24 months
  Score assessment of Becks Depression Inventory sacle

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (2):
- France (2):
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - Chu Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided